CLINICAL TRIAL: NCT04397939
Title: Association of Early Myocardial Injury With Major Adverse Outcomes in Patients With COVID-19
Brief Title: Myocardial Injury and Major Adverse Outcomes in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Annapoorna Kini, Director, Catheterization Laboratory, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 20-0965
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Myocardial Reperfusion Injury; Cardiovascular Diseases
Keywords: COVID-19; Myocardial Injury; Cardiovascular Disease; Cardiac Troponin
MeSH Terms: conditions — COVID-19; Myocardial Reperfusion Injury; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Acute Cardiac Injury: Patients with acute cardiac injury
- Patients without cardiac injury: Patients without cardiac injury
- Patients with Chronic Cardiac Injury: Patients with chronic cardiac injury

SUMMARY:
The study will analyze the incidence, clinical outcomes and predictors of myocardial injury in a large patient population with COVID-19 treated in Mount Sinai Hospital (MSH) system. In addition, the study team will explore the association between high-sensitivity troponin I (TnI) levels and clinical characteristics, biomarkers, cardiac tests data and treatment approaches to uncover the potential mechanisms responsible for COVID-19 induced myocardial injury.

DETAILED DESCRIPTION:
The study team's understanding of diagnosis, treatment and outcomes of coronavirus disease 2019 (COVID-19) is rapidly evolving. First reports from China clearly indicate that older patients with underlying cardiovascular disease and/or cardiac risk factors demonstrate higher mortality rates. Most recent reports provided novel insights into the incidence of myocardial injury in COVID-19 patients and its association with adverse outcomes. In both studies, patients with myocardial injury manifested by elevated high-sensitivity troponin I (TnI) levels had significantly higher in-hospital mortality rates compared with those without myocardial injury, (59.6 and 8.9% (3) and 51 vs 4.5 %). Among patients with myocardial injury, higher levels of TnI were associated with higher mortality rates. While the highest mortality rates were observed in patients with elevated TnI and underlying cardiovascular disease (CVD), mortality rates were also considerable in patients with elevated TnI and without prior CVD. In contrast, patients with known cardiovascular disease without TnI elevation had more favorable outcomes. Cardiac injury was independently associated with an increased risk of mortality in patients with COVID-19. The arming reports clearly indicate that the data from larger populations from multiple centers are needed to further characterize and better understand the association between myocardial injury and adverse outcomes in COVID-19 patients.

II. STUDY AIM The aim of the proposed study is to analyze the incidence, clinical outcomes and predictors of myocardial injury in a large patient population with COVID-19 treated in Mount Sinai Hospital (MSH) system. In addition, the study team will explore the association between TnI levels and clinical characteristics, biomarkers, cardiac tests data and treatment approaches to uncover the potential mechanisms responsible for COVID-19 induced myocardial injury.

III. STUDY POPULATION By October 2020, there have been 4,695 COVID-19 positive patients treated in the Mount Sinai Hospital (MSH) and more than 1,1000 patients with COVID-19 had been healed and discharged. All consecutive patients admitted to the MSH system from February 2020 to October 2020 with laboratory-confirmed COVID-19 will be included in the retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed COVID-19

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients admitted to the MSH system from February 2020 to October 2020 with laboratory-confirmed COVID-19 will be included in the retrospective study
Sampling Method: Non-Probability Sample
Enrollment: 4695 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Result] Kini A, Cao D, Nardin M, Sartori S, Zhang Z, Pivato CA, Chiarito M, Nicolas J, Vengrenyuk Y, Krishnamoorthy P, Sharma SK, Dangas G, Fuster V, Mehran R. Types of myocardial injury and mid-term outcomes in patients with COVID-19. Eur Heart J Qual Care Clin Outcomes. 2021 Sep 16;7(5):438-446. doi: 10.1093/ehjqcco/qcab053. PMID 34458912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with laboratory-confirmed COVID-19 who had a hospital encounter within the Mount Sinai Health System (New York City) between 27 February 2020 and 15 October 2020 were evaluated for inclusion.
Groups:
- Patients Without Cardiac Injury: If cardiac troponin was normal on first assessment and subsequently elevated with ≤50% variation, patients were considered as not having a myocardial injury
- Patients With Chronic Myocardial Injury: Chronic myocardial injury was considered if cardiac troponin was elevated on both first and subsequent assessments with ≤20% variation
- Patients With Acute Cardiac Injury: Acute myocardial injury was considered if (i) cardiac troponin was normal on first assessment and subsequently elevated with >50% variation, or (ii) cardiac troponin was elevated on both first and subsequent assessments with >20% variation
Period: Overall Study
Arm/Group | Patients Without Cardiac Injury | Patients With Chronic Myocardial Injury | Patients With Acute Cardiac Injury
Started | 3208 | 319 | 1168
Completed | 3208 | 319 | 1168
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Without Cardiac Injury | Patients With Chronic Myocardial Injury | Patients With Acute Cardiac Injury | Total
Number analyzed (Participants) | 3208 | 319 | 1168 | 4695
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (16.2) | 74.1 (13.5) | 72.6 (14.2) | 64.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1441 | 130 | 481 | 2052
  Male | 1767 | 189 | 687 | 2643
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 675 | 69 | 307 | 1051
  African American | 748 | 114 | 327 | 1189
  Hispanic | 1013 | 80 | 268 | 1361
  Asian | 160 | 10 | 54 | 224
  Other | 470 | 45 | 172 | 687
  Unknown | 142 | 1 | 40 | 183
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (7.2) | 27.3 (6.4) | 28.3 (7.9) | 28.9 (7.3)
Smoking, active/former [Count of Participants; unit: Participants] | 749 | 98 | 319 | 1166
Asthma [Count of Participants; unit: Participants] | 171 | 14 | 41 | 226
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 91 | 22 | 61 | 174
Hypertension [Count of Participants; unit: Participants] | 932 | 155 | 526 | 1613
Diabetes [Count of Participants; unit: Participants] | 590 | 104 | 339 | 1033
Chronic kidney disease [Count of Participants; unit: Participants] | 145 | 88 | 212 | 445
Coronary artery disease [Count of Participants; unit: Participants] | 251 | 83 | 266 | 600
Atrial fibrillation [Count of Participants; unit: Participants] | 135 | 40 | 155 | 330
Heart failure [Count of Participants; unit: Participants] | 113 | 71 | 160 | 344
Fever (T > 38.0°C) [Count of Participants; unit: Participants] | 610 | 49 | 194 | 853
Tachycardia (>100 beats/min) [Count of Participants; unit: Participants] | 1207 | 94 | 474 | 1775
Tachypnoea (≥22 breaths/min) [Count of Participants; unit: Participants] | 679 | 102 | 461 | 1242
Hypotension (Systolic Blood Pressure < 100 mmHg) [Count of Participants; unit: Participants] | 139 | 38 | 117 | 294
O2 saturation [Median (Inter-Quartile Range); unit: percent] | 91.0 [87.0 to 94.0] | 88.0 [79.0 to 91.0] | 86.0 [74.0 to 91.0] | 90.0 [83.0 to 93.0]
White blood cell count [Median (Inter-Quartile Range); unit: 10^3 cells/μL] | 7.0 [5.2 to 9.4] | 7.6 [5.4 to 10.9] | 8.5 [6.1 to 12.0] | 7.4 [5.4 to 10.2]
Neutrophil [Median (Inter-Quartile Range); unit: percent of cells] | 77.4 [67.9 to 84.2] | 80.0 [70.0 to 86.7] | 81.4 [72.8 to 87.7] | 78.6 [69.0 to 85.4]
Lymphocyte [Median (Inter-Quartile Range); unit: percent of cells] | 14.3 [9.3 to 21.7] | 12.9 [7.7 to 19.8] | 10.2 [6.5 to 16.9] | 13.3 [8.3 to 20.4]
Haemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 13.3 [12.0 to 14.4] | 12.4 [11.0 to 14.1] | 12.7 [11.0 to 14.2] | 13.1 [11.7 to 14.4]
Platelet [Median (Inter-Quartile Range); unit: 10^3 cells/μL] | 210.0 [164.0 to 274.0] | 174.0 [135.0 to 231.0] | 204.0 [154.0 to 275.5] | 206.0 [159.0 to 272.0]
C-reactive protein [Median (Inter-Quartile Range); unit: mg/L] | 95.4 [41.6 to 171.5] | 108.3 [54.3 to 184.9] | 136.9 [66.5 to 227.4] | 106.5 [48.9 to 189.0]
D-dimer [Median (Inter-Quartile Range); unit: μg/mL] | 1.2 [0.7 to 2.3] | 2.6 [1.4 to 6.6] | 2.5 [1.3 to 5.8] | 1.5 [0.8 to 3.1]
Ferritin [Median (Inter-Quartile Range); unit: ng/mL] | 608.5 [271.0 to 1300.0] | 834.0 [361.0 to 2040.0] | 853.0 [414.0 to 2062.0] | 685.5 [305.5 to 1545.5]
Blood urea nitrogen [Median (Inter-Quartile Range); unit: mg/dL] | 14.0 [10.0 to 20.0] | 39.0 [21.0 to 66.0] | 30.0 [18.0 to 51.0] | 17.0 [11.0 to 30.0]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.9 [0.7 to 1.1] | 1.7 [1.1 to 3.9] | 1.4 [0.9 to 2.4] | 1.0 [0.8 to 1.4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Death
Description: Number of deaths at 6 months follow up
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients Without Cardiac Injury: Myocardial injury was identified by high-sensitivity cardiac troponin I levels above the 99th percentile of the upper reference limit (0.03 ng/mL) with the Abbott Architect assay.
  If cardiac troponin was normal on first assessment and subsequently elevated with ≤50% variation, patients were considered as not having a myocardial injury
Arm/Group | Patients Without Cardiac Injury | Patients With Chronic Myocardial Injury | Patients With Acute Cardiac Injury
Number analyzed (Participants) | 3208 | 319 | 1168
Participants | 417 | 137 | 552

2. Secondary Outcome: Number of Participants With Pulmonary Embolism
Description: Pulmonary embolism rate as assessed by number of participants with pulmonary embolism
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Without Cardiac Injury | Patients With Chronic Myocardial Injury | Patients With Acute Cardiac Injury
Number analyzed (Participants) | 3208 | 319 | 1168
Participants | 32 | 4 | 22

3. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: Acute injury rate as assessed by number of Participants with acute kidney injury
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Without Cardiac Injury | Patients With Chronic Myocardial Injury | Patients With Acute Cardiac Injury
Number analyzed (Participants) | 3208 | 319 | 1168
Participants | 99 | 30 | 107

4. Secondary Outcome: Number of Admissions to the Intensive Care
Description: Admission to the intensive care
Time Frame: up to 6 months
Measure: Number; unit: admissions to ICU
Arm/Group | Patients Without Cardiac Injury | Patients With Chronic Myocardial Injury | Patients With Acute Cardiac Injury
Number analyzed (Participants) | 3208 | 319 | 1168
admissions to ICU | 393 | 64 | 325

ADVERSE EVENTS:
Time Frame: 6 months
Description: Retrospective chart review - Only death information obtained.
Arm/Group | Patients Without Cardiac Injury | Patients With Chronic Myocardial Injury | Patients With Acute Cardiac Injury
All-Cause Mortality (participants affected / at risk) | 417/3208 | 137/319 | 552/1168
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The time of being diagnosed as COVID-19 might not reflect the time of being infected. Troponin was not systematically assessed in all patients with COVID-19 referred to our health system, with the consequent risk of selection bias and possible overestimation of the burden of myocardial injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04397939/Prot_SAP_000.pdf